CLINICAL TRIAL: NCT05034692
Title: Application of Overlap Method to Digestive Tract Reconstruction of Totally Laparoscopic Left Colectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K202012-10
Record Dates: First submitted 2021-02-06; First posted 2021-09-05 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Colon Neoplasm
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Overlap group (Experimental): Total laparoscopic with intracorporeal anastomosis by overlap method
  Interventions: Procedure: Total laparoscopic with intracorporeal anastomosis by overlap method
- Traditional group (Active Comparator): Laparoscopic-assisted colectomy with extracorporeal anastomosis
  Interventions: Procedure: Laparoscopic-assisted colectomy with extracorporeal anastomosis

INTERVENTIONS:
Procedure: Total laparoscopic with intracorporeal anastomosis by overlap method — After the intestinal canal was dissociated and vascularized, the intestinal canal was nuded and cut off, and the distal and proximal intestinal canals were overlapped by 6 cm
  Arms: Overlap group
Procedure: Laparoscopic-assisted colectomy with extracorporeal anastomosis — After the corresponding colon and blood vessels were dissociated and treated, the carbon dioxide pneumoperitoneum was removed. The appropriate length of the incision was cut at the corresponding position of the abdomen, and the incision protector was placed. The tumor was lifted together with the free intestinal canal to the outside of the abdomen. The intestinal canals at the quasi-dismembered sites on both sides of the tumor were nuded, and the colon-colon functional end-to-end anastomosis was performed.
  Arms: Traditional group

SUMMARY:
Objective:The comparison between total laparoscopic colectomy with intracorporeal anastomosis by overlap method and laparoscopic-assisted colectomy with extracorporeal anastomosis for colon cancer surgery.

Condition or disease：Left colon cancer Intervention/treatment： Procedure:Intracorporeal left colectomy Overlap anastomosis Procedure: Extracorporeal left colectomy convention anastomosis

DETAILED DESCRIPTION:
This a simple randomized, single-center, single-blind, randomized controlled trial study.The patients were randomly divided into experimental groups and control groups by computer.The perioperative recovery data, complications and oncology index of total laparoscopic colectomy with intracorporeal anastomosis and laparoscopic-assisted colectomy with extracorporeal anastomosis would be compared.

ELIGIBILITY:
Inclusion Criteria:

* ASA<3 classification
* 18kg/m2≤BMI≤30kg/m2
* Neoplasm staging is T1-4a, N0-2, M0
* No previous history of abdominal surgery
* No previous history of neoplasm chemoradiotherapy
* No status of ileus, bowel obstruction and active hemorrhage of the digestive tract

Exclusion Criteria:

* Age<18 years or >75 years
* ASA≥3 classification
* BMI<18kg/m2 or BMI>30kg/m2
* Neoplasm staging is T4b or M1 Underwent chemoradiotherapy Appeared status of ileus,bowel perforation or active hemorrhage of digestive tract Patients with pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of early complications | one month after surgery
  According to Clavein Dindo grading standards（The scale is divided into four levels, with the minimum（Ⅰ） and the maximum（Ⅳ） level. The higher the level that more severe symptoms.）, the incidence of complications within one month after surgery, such as incision infection, bleeding, anastomotic leakage, ileus, etc., was counted

SECONDARY OUTCOMES:
anastomotic orifice stricture and torsion | one month after surgery
  According to results of intestinal barium contrast, colonoscopy and clinical symptoms to judgment
the time of first flatus | one month after surgery
  Observation of patients exhaust on days after operation
the time of first defecation | one month after surgery
  Observation of patients bowl movement on days after operation
the time of first oral feeding | one month after surgery
  Observation of patients oral intake on days after operation
postoperative hospitalization days | one month after surgery
  Observation of patients hospitalization duration on days post-surgery
the incision length and cosmetic | one month after surgery
  Comparing length and cosmetic of two groups measuring with metric
pain score | postoperative 6 hours, the first day and the third day
  Estimate for pain of subject By Visual Analog Scale for Pain (VAS Pain，The scale is divided into four levels, with the minimum（1 score） and the maximum（10 score） level. The higher the level that more severe pain.)

CONTACTS AND LOCATIONS:
Overall Officials: Wang Nan, Doctor, Study Chair — General surgery ,Tang Du of Fourth Military Medical University
Locations (1):
- General Surgery Gastrointestinal Department，Tang-Du of Fourth Military Medical University, Xi'an, Shaanxi, China